CLINICAL TRIAL: NCT06587750
Title: Cognitive Multisensory Rehabilitation, a Novel Sensorimotor Intervention for Pain Reduction in Complex Regional Pain Syndrome: a Feasibility Study
Brief Title: Cognitive Multisensory Rehabilitation for CRPS Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CharFund Jan2022 MPB
Record Dates: First submitted 2024-08-13; First posted 2024-09-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Complex Regional Pain Syndrome; CRPS; Occupational Therapy; Physiotherapy; Physical Therapy
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMR intervention (Experimental): Participants receive CMR intervention delivered by a treatment partner in a home enviornment
  Interventions: Behavioral: Cognitive Multisensory Rehabilitation

INTERVENTIONS:
Behavioral: Cognitive Multisensory Rehabilitation — CMR targets somatosensory and multisensory and cognitive functions through sensory discrimination exercises.
  Other Names: CMR

SUMMARY:
Pain treatment for Complex Regional Pain Syndrome (CRPS) is challenging. There is some evidence that pain can be reduced by therapies aimed at helping patients 'find' normal sensation in the painful body part (i.e. perceiving the exact location of a touch on the painful hand with eyes closed). In this study, a collaboration between the CRPS service at Royal United Hospital (RUH), University of the West of England (UWE), University of Bath (UoB) and Cognitive Multisensory Rehabilitation Center, the investigators aim to test whether it is possible to administer a treatment called Cognitive Multisensory Rehabilitation (CMR) to people with CRPS. In order to do this, treatment-partners (e.g. spouses, partners) will be trained to deliver CMR in a home-based environment under the supervision of a CMR specialist. Generally speaking, CMR is a rehabilitation technique in which patients are guided to better feel their painful limb by paying more attention to different sensations (e.g. touch, or position), and mindfully moving it. Since previously CMR has shown promising results in people with stroke, the investigators believe that this method could be very useful for treating pain in CRPS.

DETAILED DESCRIPTION:
Introduction This protocol describes a study aimed to investigate the feasibility and appropriateness of a novel sensorimotor treatment approach called Cognitive Multisensory Rehabilitation (CMR) for symptom reduction in people living with Complex Regional Pain Syndrome (CRPS). This study has been informed by the findings of a CRPS-patient focus group as well as clinical observations at the Royal United Hospital in Bath. The findings from this feasibility study will inform the design of larger studies to investigate the effectiveness of CMR in CRPS, offering a novel, non-drug related treatment to CRPS treatment.

Background CRPS is a chronic pain condition of unknown aetiology that commonly occurs following trauma to a limb, although it may occur spontaneously. It is defined as type 1 or type 2, depending on whether known major nerve damage is absent or present, respectively. Patients with Complex Regional Pain Syndrome commonly describe a diverse range of sensory and motor abnormalities. Sensory problems include pain to touch or the threat of touch, evoked pain, pain hypersensitivity (allodynia or/and hyperalgesia; pain due to a stimulus that does not normally provoke pain and an increased sensitivity to feeling pain and an extreme response to pain, respectively), but at the same time non-noxious sensory loss (hypoesthesia). Motor problems include troubles in initiating movement, weakness and reduced function amongst others.

Clinical features often present in people living with CRPS commonly resulting in patients having difficulty to engage with their affected limb and therefore having a detrimental effect on rehabilitation outcomes are:

* Body perception disturbances: the reported individual's perceived alteration of their CRPS affected body part while regarding the remainder of their body as normal.
* Loss of self-ownership and amputation desire: patients' perception that the painful limb(s) do not belong to them and the desire to amputate these body parts.
* Allodynia: painful response to a stimulus that does not normally produce pain.
* Motor impairments: including tremor, decreased range of movement, muscle weakness, and/or having the affected limb set in a sustained, fixed posture (i.e. dystonia).

Sensorimotor interventions (i.e. interventions aiming to improve sensory and motor feedback of the affected limb) have shown promising outcomes on increasing perception associated with the affected limb (i.e. tactile acuity; precision with which we can sense touch) and decreasing pain intensity. Although its mechanisms are largely unknown, it is thought that the 'normalized' sensory and motor feedback may compete with pain stimulus resulting in pain reduction in people with CRPS. The evidence for the effectiveness of these treatment modalities in CRPS is weak, and often focus only on pain reduction. Thus further research is required on novel sensorimotor interventions that target also other abnormalities present in CRPS (i.e. body perception disturbances, loss of self-ownership and amputation desire and motor impairments).

Cognitive Multisensory Rehabilitation is a term agreed by the International Cognitive Multisensory Rehabilitation Centre to describe a sensorimotor intervention originally developed for stroke motor rehabilitation by Professor Perfetti (1940-2020). CMR targets somatosensory and multisensory and cognitive functions through sensory discrimination exercises. It focuses on the perception and integration of different sensory modalities (e.g. somatosensory, visual, etc.) and body parts (e.g. shoulder and hand) in order to produce purposeful, effective and accurate movements allowing an appropriate relationship with the surrounding environment. Clinical observations from the CRPS service at the Royal United Hospital (RUH) have suggested that CMR may have an impact on symptom reduction (e.g. decreased body perception disturbances or pain reduction) as a part of a multidisciplinary rehabilitation programme.

In contrast to other sensorimotor interventions, CMR offers a comprehensive range of sensorimotor tasks targeting a wider range of sensorimotor, cognitive and body representation impaired functions in CRPS (i.e. body perception disturbances, loss of self-ownership and amputation desire, allodynia and motor impairments). In CMR, patients are guided to increase their affected limb's perception by discriminating different sensory information through the activation of cognitive processes (such as perception, attention or body representation) and mindful movements.

Furthermore, unlike sensorimotor interventions, CMR tasks are considered to be discrimination-based: e.g. the patient has to recognise different types of stimuli on the painful limb, such as which fabric they feel (i.e. tactile discrimination). Because of this, CMR interventions require a trained facilitator whose role is to help the patients to recognise the different sensory information with eyes closed by physically guiding the patient as well as posing the cognitive question. Preliminary data has shown that improvements in pain levels observed following sensorimotor interventions were enhanced and lasted longer if people with CRPS discriminated between different stimuli as opposed to just receiving sensory stimulation on the painful body part. This suggested that a broader activation of cognitive processes such as problem solving, attention and perception may increase the effectiveness of sensorimotor interventions.

Recently, Covid-19 restrictions have prompted the increase of home-based treatment complementing therapy treatment. Home-based discrimination sensory retraining has shown promising results in pain reduction for people with CRPS.

ELIGIBILITY:
Inclusion Criteria:

* Participants meet the Budapest criteria for Type I CRPS4 (i.e. the diagnostic criteria for CRPS) in one limb (unilateral).
* Pain duration for a minimum of 3 months.
* 18 years in age or older.
* Able to understand verbal and written English.
* Willing to participate and provide written informed consent.
* Have not previously received CMR.
* Have someone available to act as treatment facilitator and consent to participate in the study.

Exclusion Criteria:

* Presence of any co-morbidity that may influence CRPS symptoms including stroke, diabetic peripheral neuropathy, progressive neurological disease such as multiple sclerosis, and Parkinson's disease.
* Presence of Post-Traumatic Stress Disorder or other psychological conditions hindering patients' ability to engage with the intervention.
* Serious ill health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Number of sessions (number of total sessions), duration (total duration of intervention in minutes), frequency (number of sessions over 4 weeks), presence of any exacerbation of symptoms (number total of symptom exacerbation). | Pre-post intervention (4 weeks)
  Suitability
Number of sessions (number of total sessions), duration (total duration of intervention in minutes), frequency (number of sessions over 4 weeks), presence of any exacerbation of symptoms (number total of symptom exacerbation). | Pre-post intervention (4 weeks)
  Feasibility

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory (ranging from 0-100, higher score indicates worse outcome) | Pre-post intervention (4 weeks)
  Pain
Tampa Scale of Kinesiophobia (ranging from 17-68, higher score indicates worse outcome) | Pre-post intervention (4 weeks)
  Kinesiophobia
The Bath CRPS body perception disturbance scale (ranging from 0-57, higher score indicate worse outcome) | Pre post intervention (4 weeks)
  Body perception disturbance of painful limb
Evaluation of Daily Activity Questionnaire (ranging from 0-147, higher scores indicate worse outcome) | Pre post intervention (4 weeks)
  Physical function
EQ-5D-5L (0-100, higher value indicates better outcome) | Pre post intervention (4 weeks)
  Quality of life
Tactile acuity (higher value indicates worse outcome) | Pre post intervention (4 weeks)
  Two point discrimination threshold at the pulp of the index finger or hallux
Numerical Rating Scale (0-10, higher outcome indicates worse outcome) | Pre post intervention (4 weeks)
  Pain

CONTACTS AND LOCATIONS:
Overall Officials: Jane Carter, Head, Study Chair — Royal United Hospital
Locations (1):
- Royal United Hospital, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT06587750/Prot_000.pdf
  • Informed Consent Form (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT06587750/ICF_001.pdf